CLINICAL TRIAL: NCT06700889
Title: Investigating the Relationship Between Glycemia and Sleep in Adults With Cystic Fibrosis-Related Diabetes
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Trustees of Dartmouth College (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Hassan Dashti, Assistant Professor, Massachusetts General Hospital
Other Study IDs: 2024P000762
Record Dates: First submitted 2024-11-18; First posted 2024-11-22 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis Related Diabetes; Hyperglycaemia; Insomnia; Cardiometabolic Diseases; Circadian Rhythm Disorders
Keywords: Cystic Fibrosis Related Diabetes; Tube Feeds; Circadian Rhythm; Diabetes; Home Enteral Nutrition; Circadian misalignment; Nutrition
MeSH Terms: conditions — Hyperglycemia; Sleep Initiation and Maintenance Disorders; Chronobiology Disorders; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HEN group: This group will include participants who habitually use home enteral nutrition (HEN).
- No HEN Group: This group will include participants who do not use home enteral nutrition (HEN).

SUMMARY:
The goal of this at-home, remote study is to understand the relationship between blood sugars and sleep in adults living with Cystic Fibrosis Related Diabetes (CFRD).

DETAILED DESCRIPTION:
The study is a 10-day home-based, observational study of 30 adults with CFRD aimed at concurrently phenotyping glucose, sleep, and circadian rhythms. The remote study is designed to reduce participant burden while allowing for safe and robust objective data and specimen collection and to inform future clinical trial design. The objective of the proposed pilot and feasibility clinical study is to assess the feasibility of remotely phenotyping glycemia, sleep, and circadian rhythms of adults living with CFRD and to generate preliminary data to power a future clinical trial.

ELIGIBILITY:
Inclusion Criteria:

Adult men or non-pregnant women volunteers (age 18-79) Able and willing to give consent and comply with procedures Known diagnosis of CF Related Diabetes (CFRD) and clinically stable with no significant changes in therapies within the prior 3 months

Concomitant Medications:

A. No initiation of an investigational drug within prior 28 days B. No initiation of new chronic therapy (e.g., ibuprofen, azithromycin, inhaled tobramycin, Cayston®) within prior 28 days C. No acute use of antibiotics (oral, inhaled or IV) or acute use of systemic corticosteroids for respiratory tract symptoms within prior 14 days D. No starting/stopping modulator therapy in the prior 3 months

Exclusion Criteria:

Blind, deaf, or unable to speak English Pregnant, nursing, or plan on pregnancy Current use of melatonin and unwilling to stop during the study With skin condition that precludes wearing sensors Within the last 4 weeks, acute CF exacerbation requiring IV antibiotics or hospitalization Major changes in diet or physical activity level in the last 4 weeks Untreated sleep and circadian disorders

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cystic fibrosis-related diabetes patients living in the US and identified from various sources: Rally website, the MGH Adult CF Program, the CF Foundation EnVision program, and the Oley Foundation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-01-08 (Actual); Study Completion 2026-01-08 (Actual)

PRIMARY OUTCOMES:
Completion Rate | 10 days
  Primary feasibility measure, defined by the completion of all study procedures and the return of study devices after the 10-day study period.

SECONDARY OUTCOMES:
Enrollment Rate | Through study completion, an average of 1 year
  Feasibility measure, assessing the number of participants who successfully enroll.
Percentage of time glucose levels | 10 days
  Percentage of time glucose levels are within 70-180 mg/dL, derived from CGM.
Number of CGM Days | 10 days
  Total number of days with usable CGM data collected across participants.
Number of Actigraphy Days | 10 days
  Total number of days with usable actigraphy data collected across participants.
Number of Completed At-Home Kits (HbA1c) | 10 days
  Total number of at-home HbA1c kits successfully completed and returned.
Total number of days with usable food records collected across participants. | 10 days
  Total number of days with usable food records collected across participants.
Percentage of Time Above Range (>180 mg/dL) | 10 days
  Percentage of time glucose levels are above 180 mg/dL, derived from CGM.
Time Below Range (<54 mg/dL) | 10 days
  Percentage of time glucose levels fall below 54 mg/dL, derived from CGM.
Mean Glucose | 10 days
  Average glucose level across the study period, derived from CGM.
Glucose Variability | 10 days
  Variability in glucose levels, including standard deviation and coefficient of variability, derived from CGM.
Number of Awakenings | 10 days
  Total number of awakenings during the sleep period, measured by actigraphy.
Wake After Sleep Onset (WASO) | 10 days
  Total time in minutes spent awake after initially falling asleep, measured by actigraphy.
Sleep Efficiency | 10 days
  Ratio of sleep duration to time in bed, expressed as a percentage, measured by actigraphy.
Sleep Latency | 10 days
  Time taken to fall asleep after going to bed, measured by actigraphy.
Intradaily Stability | 10 days
  A measure of consistency in daily activity patterns, derived from actigraphy.
Interdaily Variability | 10 days
  A measure of day-to-day variability in activity patterns, derived from actigraphy.
Daily Energy Intake | 4 days
  Total daily caloric intake derived from food records.
Healthy Eating Index | 4 days
  Indicator of dietary quality derived from food records.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan S Dashti, Ph.D., R.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share Individual Participant Data (IPD) with other researchers as the information collected, which includes detailed glucose profiles, sleep patterns, and circadian rhythm data from individuals with CFRD, is classified as protected health information.

REFERENCES:
- See also: Rally | Cystic Fibrosis Related Diabetes and Tube Feeding — https://rally.massgeneralbrigham.org/study/cfrd_tubefeed